CLINICAL TRIAL: NCT04686201
Title: Development of Diabetes Mobile Application "MyD App" To Improve Patient's Knowledge, Compliance and Control: An Interventional Study Among Uncontrolled Type 2 Diabetes Mellitus Patients in Kedah, Malaysia
Brief Title: Development of Diabetes Mobile Application
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Diabetes Apps
Record Dates: First submitted 2020-12-20; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Device: Diabetes Mobile Application
- control group (No Intervention)

INTERVENTIONS:
Device: Diabetes Mobile Application — incorporating mobile application usage in managing diabetes mellitus patient in health clinics
  Arms: intervention group

SUMMARY:
this study is to measure the effectiveness of a diabetes mobile application for improving patient's knowledge, compliance and diabetes control among uncontrolled Type 2 Diabetes Mellitus mellitus patients in Kedah

DETAILED DESCRIPTION:
Specific Objective

1. To develop and validate a diabetes mobile-app (MyD-App) for patients with uncontrolled Type 2 Diabetes Mellitus.
2. To measure the effectiveness of a diabetes mobile application for improving knowledge, compliance and control using the newly developed and validated MyD-App among patients with uncontrolled Type 2 Diabetes Mellitus.

Hypothesis

1. There is an increased in patient's knowledge on diabetes after MyD-App usage.
2. There is an increased in patient's compliance on medication and treatment after MyD-App usage.
3. There is a diabetes control improvement (HbA1C < 6.5% or HbA1C reduction ≥ 1%) among Type 2 Diabetes Mellitus patients in Kedah after MyD-App usage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Diagnosed with type 2 diabetes mellitus by a registered medical doctor.
* Registered and actively follow up in the health clinics at selected districts. (actively follow up: follow up at the clinic for at least once in a year).
* Own a smartphone with the Android platform.
* HbA1C >7%

Exclusion Criteria:

* GDM
* Illiterate
* Anemia / Thalassemia
* Not agree to be the sample for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of uncontrolled Diabetes Mellitus patients who have good knowledge after using Diabetes Mobile Application | 6 months
  Percentage of uncontrolled Diabetes Mellitus patients who have good knowledge after using Diabetes Mobile Application (assessment using Michigan Diabetes Knowledge Test Questionnaire)
Percentage of uncontrolled Diabetes Mellitus patients who have good compliance after using Diabetes Mobile Application | 6 months
  Percentage of uncontrolled Diabetes Mellitus patients who have good compliance after using Diabetes Mobile Application (assessment using Malaysia Medication Adherence Assessment Tool (MyMAAT) for diabetic patients)
Percentage of uncontrolled Diabetes Mellitus patients who have good control diabetes after using Diabetes Mobile Application | 6 months
  Percentage of uncontrolled Diabetes Mellitus patients who have good control diabetes (HbA1C 7% or more than 1% reduction of HbA1C) after using Diabetes Mobile Application

CONTACTS AND LOCATIONS:
Overall Officials: MOHD ROHAIZAT HASSAN, PhD, Principal Investigator — Department of Community Health, Faculty of Medicine, Universiti Kebangsaan Malaysia
Locations (1):
- Jabatan Kesihatan Negeri Kedah, Alor Star, Kedah, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided